CLINICAL TRIAL: NCT06043518
Title: Functional, Structural, and Metabolic Central Nervous System Changes Following Damage of the Central Nervous System
Brief Title: CNS Changes Following Upper Limb Loss
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00937 - Upper Limb Loss
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Amputation, Congenital; Upper Limb; Amelia
Keywords: Plasticity; Congenital amputee; Upper limb amelia; Somatotopy; Functional MRI; Hand; Reorganisation
MeSH Terms: conditions — Amputation, Congenital; Ectromelia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with congenital amputation
  Interventions: Diagnostic Test: MRI
- Healthy subjects
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Use of functional and structural MRI in both the brain and the spinal cord as well as questionnaires and clinical measures of motor function
  Groups: Patients with congenital amputation
Diagnostic Test: MRI — Use of functional and structural MRI in both the brain and the spinal cord and questionnaires.
  Groups: Healthy subjects

SUMMARY:
The objective of this study is to better understand the structural and functional changes that the central nervous system (CNS) undergoes following congenital upper limb loss. The focus is on the brain's sensory processing and how neuronal changes may relate to clinical measures. By doing so, the hope is to gain insight into the contribution of critical periods to the plasticity of the sensorimotor processing stream. Both macroscopic and microscopic changes of the brain will be examined in individuals with upper limb amelia and compared to healthy controls. fMRI will be combined with behavioural testing to understand which clinical and behavioural determinants drive somatosensory representations along the entire somatosensory processing stream. Using advanced imaging techniques, the aim is to investigate the contribution of brainstem reorganisation to plasticity observed at the cortical level and, by doing so, gain a better understanding of the mechanistic underpinnings of functional reorganisation. Overall, the hope is to provide the first mechanistic insight into whether early life experiences are crucial for the development of the relay nuclei in the central nervous system and how these changes relate to clinical measures such as adaptive behaviours or pain.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Age 18-75
* Upper-limb congenital amputees with complete absence of a hand
* Signed informed consent

Exclusion Criteria - Patients:

* Contraindications to magnetic resonance imaging
* Neurological impairment of body function impairments not induced by spinal cord injury
* BMI > 40
* Pregnancy
* Claustrophobia

Inclusion Criteria - Healthy subjects:

* Age 18-75
* Signed Informed consent

Exclusion Criteria - Healthy subjects:

* Contraindications to magnetic resonance imaging
* Pregnancy
* Neurological illness
* Impairment of body function induced by a congenital upper-limb amputation
* Claustrophobia
* BMI > 40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an upper-limb amputation and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of functional MRI (fMRI) parameter between 2 to 4 time points | Up to 50 weeks
  Change of brain activities is assessed between 2 to 4 time points using fMRI during resting-state or a specific task in patients with congenital amputations and compared to healthy controls

SECONDARY OUTCOMES:
Conventional magnetic resonance imaging (MRI) parameter | Up to 50 weeks
  Structural characteristics in the brain and cervical spinal cord are assessed in patients with congenital upper-limb amputations using conventional MRI and compared to healthy controls
Amputees: Motor Activity Log questionnaire | Up to 50 weeks
  Evaluation of residual limb and/or prosthesis usage as compared to other body parts via a questionnaire and behavioural assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof., Principal Investigator — University of Zurich
Locations (1):
- Balgrist Campus, Zurich, Canton of Zurich, Switzerland